CLINICAL TRIAL: NCT02992574
Title: Post-Mastectomy Radiation Therapy in High Risk, Node Negative Women With Early Breast Cancer (PMRT-NNBC)
Brief Title: Trial Evaluating Role of Post Mastectomy Radiotherapy in Women With Node Negative Early Breast Cancer
Acronym: PMRT-NNBC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Principal Investigator, Dr. Tabassum Wadasadawala, Associate Professor, Radiation Oncology, Tata Memorial Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1602; CTRI/2016/12/007532 (Registry Identifier: Clinical Trial Registry- India)
Record Dates: First submitted 2016-12-11; First posted 2016-12-14 (Estimated); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Breastcancer
Keywords: Post-Mastectomy Radiation; Node Negative; Early breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Arm Experimental Post Mastectomy Radiotherapy Arm No Intervention: No Post Mastectomy Radiotherapy
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Post Mastectomy Radiation Therapy (PMRT) (Experimental): Post mastectomy radiotherapy will be given
  Interventions: Radiation: Post Mastectomy Radiation therapy
- Observation (No PMRT) (No Intervention): No adjuvant radiotherapy will be given.

INTERVENTIONS:
Radiation: Post Mastectomy Radiation therapy — Post mastectomy radiotherapy to the chest wall and ipsilateral supra-clavicular fossa to a dose of 40 Gy in 15 fractions over 3 weeks
  Other Names: PMRT
  Arms: Post Mastectomy Radiation Therapy (PMRT)

SUMMARY:
Postmastectomy radiotherapy (PMRT) is unequivocally beneficial in reducing the recurrences as well as improving survival in node positive breast cancer patients. PMRT for women with T1-T2 tumors and negative axillary nodes is not generally warranted because of the presumed low risk of recurrence in this population as a whole. However, in the setting of multiple adverse prognostic factors, the recurrence risk approaches and in some cases surpasses the risk of recurrence documented for patients with one to three positive lymph nodes. Numerous retrospective series have reported the outcome and patterns of failure for post-mastectomy patients treated without radiation. Many of these series have analyzed several high risk factors which were predictive of loco-regional recurrence wherein the role of adjuvant post-mastectomy radiation can be considered. Some authors have used combinations of prognostic factors, such as age, tumour size, grade, receptor status, Her2neu status and lympho-vascular space invasion to define subgroups with more specific risks of loco-regional recurrence than single factors alone. The current trial hypothesizes that "Post-mastectomy radiation in high risk, node negative early breast cancer patients decreases rates of loco-regional recurrence and improves disease free survival" and propose to address the question in randomized setting.

ELIGIBILITY:
Inclusion Criteria:

* Women with unilateral pT1,2N0M0 breast cancer or multifocal breast cancer if largest discrete tumour at least 2cm or if the tumour area comprises multiple small adjacent foci of invasive carcinoma then overall maximum dimension taken. This must be greater than 2cm.
* Upfront total mastectomy (with minimum 1 mm margin clear of invasive cancer or DCIS) and axillary staging procedure (clearance, sampling or SNB)
* T2 tumors with one risk factor or T1 tumors with any of the following two high risk factors such as presence of high grade, lymphovascular invasion, ER/PR negative, HER2 positivity, age < 35 years.
* Fit to receive adjuvant radiation +/- chemotherapy (if indicated) +/- hormonal therapy (if indicated)
* Written, informed consent

Exclusion Criteria:

* Any pTis/3/4, M1 patients
* Patients who have any pathologically involved axillary nodes (micro-metastasis may be allowed)
* Patients who have undergone neoadjuvant systemic therapy.
* Previous or concurrent malignancy other than non melanomatous skin cancer and carcinoma in situ of the cervix
* Pregnancy
* Bilateral breast cancer
* Not fit for surgery, radiotherapy or adjuvant systemic therapy
* Unable or unwilling to give informed consent

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1022 (Estimated)
Dates: Start 2016-05-27 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 5 years
  This will be measured using Kaplan Meier time to event analysis

SECONDARY OUTCOMES:
Chest wall recurrence | 5 years
  This is the incidence of local recurrence in the chest wall
Regional recurrence | 5 years
  This is the incidence of recurrence in the regional lymphatics
Metastasis-free survival | 5 years
  This will be measured using Kaplan Meier time to event analysis
Overall survival | 5 years
  This will be measured using Kaplan Meier time to event analysis
Acute Morbidity of radiotherapy | 4 weeks from the start of radiotherapy
  RTOG Acute radiation morbidity scoring
Late Morbidity of radiotherapy | 6 months from end of radiotherapy to 5 years
  RTOG Late radiation morbidity scoring
Quality of life scores under different domains of the QLQ C-30 and BR-23 questionnaires | 5 years post surgery
  Quality of life will be assesses by EORTC QLQ C-30 core questionnaire and the breast cancer specific module BR-23 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Tabassum Wadasadawala, MBBS,MD,DNB, Principal Investigator — Assistant Professor, Radiation Oncology, Tata Memorial Centre
Locations (7):
- India (7):
  - Post Graduate Institute of Medical Education & Research, Chandigarh, Chandigarh
  - Kolhapur Cancer Centre Pvt Ltd, Kolhāpur, Maharashtra
  - Tata Memorial Centre, Mumbai, Maharashtra
  - Max Super Speciality Hospital, Shalimar Bagh, Delhi, National Capital Territory of Delhi
  - Max Super Speciality Hospital(A unit of Devki Devi Foundation), New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Bhagwan Mahaveer Cancer Hospital and Research Centre, Jaipur, Rajasthan

IPD SHARING:
Plan to Share IPD: No